CLINICAL TRIAL: NCT06028438
Title: A Phase 2a Multicenter, Randomized, Double Blind, Parallel, Proof of Concept Study Evaluating the Efficacy and Safety of Nipocalimab and Certolizumab Combination Therapy in Participants With Active Rheumatoid Arthritis Despite Prior Treatment With Advanced Therapies (bDMARD or tsDMARD)
Brief Title: A Study to Evaluate the Nipocalimab and Certolizumab Combination Therapy in Participants With Active Rheumatoid Arthritis
Acronym: DAISY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109343; 2023-504045-31-00 (Registry Identifier: EUCT number); 80202135ARA2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Certolizumab + Placebo (Active Comparator): Participants will receive placebo intravenously (IV) and certolizumab dose 1 subcutaneously at Week 0, 2, and 4 followed by placebo IV and certolizumab dose 2 subcutaneously at Weeks 6 to 22.
  Interventions: Drug: Placebo; Drug: Certolizumab
- Certolizumab + Nipocalimab (Experimental): Participants will receive nipocalimab IV and certolizumab dose 1 subcutaneously at Week 0, 2, and 4 followed by nipocalimab IV and certolizumab dose 2 subcutaneously at Weeks 6 to 22.
  Interventions: Drug: Nipocalimab; Drug: Certolizumab

INTERVENTIONS:
Drug: Placebo — Placebo will be administered intravenously.
  Arms: Certolizumab + Placebo
Drug: Nipocalimab — Nipocalimab will be administered intravenously.
  Other Names: JNJ-80202135; M281
  Arms: Certolizumab + Nipocalimab
Drug: Certolizumab — Certolizumab will be administered subcutaneously.
  Other Names: Cimzia

SUMMARY:
The purpose of this study is to evaluate the efficacy of combination therapy with nipocalimab and certolizumab compared to certolizumab monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) and meeting the 2010 American college of rheumatology (ACR) or European League Against Rheumatism (EULAR) criteria for RA for at least 3 months before screening
* Has moderate to severe active RA as defined by persistent disease activity with at least 6 of 66 swollen joints and 6 of 68 tender joints at the time of screening and at baseline
* Is positive for anti-citrullinated protein antibodies (ACPA) or rheumatoid factor (RF) by the central laboratory at the time of screening
* Has C-reactive protein (CRP) greater than or equal to (>=) 0.3 milligram per deciliter (mg/dL) by the central laboratory at the time of screening
* If has received prior biological disease-modifying antirheumatic drugs (bDMARDs) (or biosimilars) other than anti-tumor necrosis factor (anti-TNF) agent in RA, has demonstrated inadequate response (IR) or intolerance to the therapy based on one of the following:

  1. IR to at least 1bDMARD (or the biosimilars) other than anti-TNF agents, as assessed by the treating physician, after at least 12 weeks of therapy including but not limited to abatacept, anakinra, tocilizumab, and sarilumab or at least 16 weeks of therapy with rituximab Documented IR may include inadequate improvement or loss in response after initial improvement in joint counts or other parameters of disease activity
  2. Intolerance to bDMARD (or biosimilars) other than anti-TNF agent, as assessed by the treating physician. Documented intolerance includes side effects and injection or infusion reactions
* If has received prior anti-TNF agent (including biosimilars), has demonstrated IR to >=1 anti-TNF agent (including biosimilars), as assessed by the treating physician:

  1. After at least 12 weeks dosage of etanercept, adalimumab, golimumab (including biosimilars), and/or
  2. After at least 14 weeks dosage (example, at least 4 doses) of infliximab (including biosimilars) Documented IR may include inadequate improvement or loss in response after initial improvement in joint counts or other parameters of disease activity

Exclusion Criteria:

* Has a confirmed or suspected clinical immunodeficiency syndrome not related to treatment of RA or has a family history of congenital or hereditary immunodeficiency unless confirmed absent
* Is (anatomically or functionally) asplenic
* Has experienced myocardial infarction, unstable ischemic heart disease, or stroke less than or equal to (<=) 12 weeks of screening
* Has a diagnosis of congestive heart failure including medically controlled, asymptomatic congestive heart failure
* Has a history of known demyelinating disease such as multiple sclerosis or optic neuritis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (32):
- United States (10):
  - Arizona Arthritis and Rheumatology Research PLLC, Phoenix, Arizona
  - Newport Huntington Medical Group, Huntington Beach, California
  - Inland Rheumatology Clinical Trials Inc., Upland, California
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Integral Rheumatology And Immunology Specialists, Plantation, Florida
  - Atlanta Research Center for Rheumatology, Marietta, Georgia
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Southwest Rheumatology Research LLC, Mesquite, Texas
- Argentina (7):
  - STAT Research S A, Buenos Aires
  - Centro Privado de Medicina Familiar, Buenos Aires
  - Sanatorio Agote, Buenos Aires
  - Hospital Central Militar Cirujano Mayor Dr Cosme Argerich, Buenos Aires
  - Mautalen Salud e Investigacion, CABA
  - ARCIS Salud SRL Aprillus asistencia e investigacion, CABA
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán
- Germany (3):
  - Hamburger Rheuma Forschungszentrum II, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Rheumazentrum Ratingen, Ratingen
- Hungary (5):
  - Budai Irgalmasrendi Korhaz, Budapest
  - Bekes Varmegyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Porcika Klinika - Vasarhelyi Sarkanyfu Kft., Hódmezővásárhely
  - CMed Rehabilitacios es Diagnosztikai Kozpont, Székesfehérvár
  - Vital Medical Center Orvosi es Fogaszati Kozpont, Veszprém
- Poland (4):
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - NZOZ Lecznica MAK MED S C, Nadarzyn
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Centrum Medyczne Reuma Park, Warsaw
- United Kingdom (3):
  - Western General Hospital, Edinburgh
  - Medway NHS Foundation Trust, Gillingham
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical- trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Certolizumab and Placebo: Participants received certolizumab 400 milligram (mg) subcutaneously (SC) at Weeks 0, 2, and 4 followed by certolizumab 200 mg SC every 2 weeks (q2w) from Week 6 up to Week 22 and placebo matching to nipocalimab intravenously (IV) q2w starting from Week 0 up to Week 22.
- Group 2: Certolizumab and Nipocalimab: Participants received nipocalimab 30 milligrams per kilogram (mg/kg) IV q2w starting from Week 0 up to Week 22 and certolizumab 400 mg SC at Weeks 0, 2, and 4 followed by certolizumab 200 mg SC q2w from Week 6 up to Week 22.
Period: Overall Study
Arm/Group | Group 1: Certolizumab and Placebo | Group 2: Certolizumab and Nipocalimab
Started | 41 | 62
Completed | 32 | 49
Not Completed | 9 | 13
Not completed — Adverse Event | 3 | 9
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Certolizumab and Placebo: Participants received certolizumab 400 mg SC at Weeks 0, 2, and 4 followed by certolizumab 200 mg SC q2w from Week 6 up to Week 22 and placebo matching to nipocalimab IV q2w starting from Week 0 up to Week 22.
- Group 2: Certolizumab and Nipocalimab: Participants received nipocalimab 30 mg/kg IV q2w starting from Week 0 up to Week 22 and certolizumab 400 mg SC at Weeks 0, 2, and 4 followed by certolizumab 200 mg SC q2w from Week 6 up to Week 22.
- Total: Total of all reporting groups
Arm/Group | Group 1: Certolizumab and Placebo | Group 2: Certolizumab and Nipocalimab | Total
Number analyzed (Participants) | 41 | 62 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 53 | 89
  >=65 years | 5 | 9 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (9.49) | 55 (8.96) | 53.8 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 57 | 91
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 20 | 37
  Not Hispanic or Latino | 24 | 42 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 37 | 56 | 93
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 9 | 15 | 24
  Germany | 4 | 5 | 9
  Hungary | 5 | 12 | 17
  Poland | 8 | 12 | 20
  United Kingdom | 1 | 0 | 1
  United States | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Index Score 28 Using C-reactive Protein (DAS28-CRP) at Week 12
Description: Change from baseline in DAS28-CRP at Week 12 were reported. The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity, and C-reactive protein (CRP; in milligrams per liter [mg/L]). The set of 28 joint count was based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. Score on the DAS28 ranged from 0 to 10, where higher scores indicated more disease activity. Negative changes from baseline indicated improvement of arthritis.
Time Frame: Baseline (Week 0), Week 12
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose (partial or complete) of any study intervention.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Group 1: Certolizumab and Placebo | Group 2: Certolizumab and Nipocalimab
Number analyzed (Participants) | 41 | 62
Score on a Scale | -1.86 [-2.55 to -1.17] | -1.92 [-2.59 to -1.25]
Statistical Analysis 1: Comparison: Group 1: Certolizumab and Placebo vs Group 2: Certolizumab and Nipocalimab; Test type: Superiority; p = 0.822, ANCOVA; Least square mean difference = -0.06, 95% CI 2-sided [-0.60 to 0.48]

2. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology (ACR) Response 20 at Week 12
Description: ACR20 response is defined as: greater than or equal to (>=)20 percent (%) improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=20% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 millimeters [mm], 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function as measured by Disability Index of Health Assessment Questionnaire (HAQ-DI; 20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area), and CRP.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Certolizumab and Placebo | Group 2: Certolizumab and Nipocalimab
Number analyzed (Participants) | 41 | 62
Percentage of participants | 63.4 | 62.9

3. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology (ACR) 50 Response at Week 12
Description: Percentage of participants who achieved ACR50 at Week 12 were reported. ACR50 response is defined as: >=50% improvement from baseline in both tender joint count (68 joints) and swollen joint count (66 joints), and >=50% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function as measured by Disability Index of Health Assessment Questionnaire (HAQ-DI; 20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area), and CRP.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Certolizumab and Placebo | Group 2: Certolizumab and Nipocalimab
Number analyzed (Participants) | 41 | 62
Percentage of participants | 31.71 | 40.32

4. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology (ACR) 70 Response at Week 12
Description: Percentage of participants who achieved ACR70 response at Week 12 were reported. ACR70 response is defined as: >=70% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=70% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using VAS (0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function as measured by (HAQ-DI) 20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area), and CRP.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Certolizumab and Placebo | Group 2: Certolizumab and Nipocalimab
Number analyzed (Participants) | 41 | 62
Percentage of participants | 12.20 | 14.52

5. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology (ACR) 90 Response at Week 12
Description: Percentage of participants who achieved ACR90 response at Week 12 were reported. ACR90 response is defined as: >=90% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=90% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using VAS (0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function as measured by HAQ-DI (20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area), and CRP.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Certolizumab and Placebo | Group 2: Certolizumab and Nipocalimab
Number analyzed (Participants) | 41 | 62
Percentage of participants | 2.44 | 3.23

6. Secondary Outcome: Percentage of Participants Who Achieved Disease Activity Index Score 28 Using C-reactive Protein (DAS28-CRP) Remission at Week 12
Description: The DAS28 remission is defined as DAS28 -CRP value of less than (<) 2.6 at Week 12. The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity, and CRP (in milligrams per liter [mg/L]). The set of 28 joint count was based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. Score on the DAS28 ranged from 0 to 10, where higher scores indicated more disease activity. Negative changes from baseline indicated improvement of arthritis.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Certolizumab and Placebo | Group 2: Certolizumab and Nipocalimab
Number analyzed (Participants) | 41 | 62
Percentage of participants | 14.63 | 25.81

7. Secondary Outcome: Percentage of Participants Who Achieved Disease Activity Index Score 28 Using C-reactive Protein (DAS28-CRP) Low Disease Activity (LDA) at Week 12
Description: Percentage of participants who achieved DAS28-CRP LDA at Week 12 were reported. DAS28 LDA is defined as a DAS28 value of less than or equal to (<=3.2) at a visit. The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity, and CRP (in milligrams per liter [mg/L]). The set of 28 joint count was based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. Score on the DAS28 ranged from 0 to 10, where higher scores indicated more disease activity. Negative changes from baseline indicated improvement of arthritis.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Certolizumab and Placebo | Group 2: Certolizumab and Nipocalimab
Number analyzed (Participants) | 41 | 62
Percentage of participants | 26.83 | 43.55

8. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Week 12
Description: Change from baseline in HAQ-DI score at Week 12 were reported. The HAQ-DI is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas: dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living, over the past week. Responses in each functional area were scored on a scale from 0 (indicating no difficulty) to 3 (inability to perform a task in that area). Overall score was computed as the sum of category scores and divided by the number of categories answered, score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
Time Frame: Baseline (Week 0), Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Group 1: Certolizumab and Placebo | Group 2: Certolizumab and Nipocalimab
Number analyzed (Participants) | 41 | 62
Score on a scale | -0.33 [-0.62 to -0.04] | -0.30 [-0.58 to -0.02]

9. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score at Week 12
Description: Change from baseline in CDAI at Week 12 were reported. The CDAI score is a derived score combining 4 disease assessments: tender joint counts (28 joints), swollen joint counts (28 joints), Patient's Global Assessment of Disease Activity (PtGA), and Physician's Global Assessment of Disease Activity (PGA). Change from baseline in CDAI score measured the change in disease activity, where a negative change indicated an improvement, and a positive change indicated a worsening. The total score range is 0-76. Score interpretation: Remission <=2.8; Low Disease Activity CDAI > 2.8 and <=10; Moderate Disease Activity CDAI >10 and <=22; High Disease Activity CDAI > 22.
Time Frame: Baseline (Week 0), Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Group 1: Certolizumab and Placebo | Group 2: Certolizumab and Nipocalimab
Number analyzed (Participants) | 41 | 62
Score on a scale | -22.51 [-29.23 to -15.78] | -21.36 [-27.89 to -14.83]

ADVERSE EVENTS:
Time Frame: All-cause mortality: From screening (-6 weeks) up to Week 30; Serious and Other AEs: From Week 0 up to Week 30
Description: The safety analysis set included all randomized participants who received at least 1 dose (partial or complete) of any study intervention.
Arm/Group | Group 1: Certolizumab and Placebo | Group 2: Certolizumab and Nipocalimab
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/41 | 7/62
Other Adverse Events (participants affected / at risk) | 7/41 | 23/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Certolizumab and Placebo (N=41) | Group 2: Certolizumab and Nipocalimab (N=62)
Myocardial Infarction (Cardiac disorders) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 | 1
Soft Tissue Infection (Infections and infestations) | 1 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Certolizumab and Placebo (N=41) | Group 2: Certolizumab and Nipocalimab (N=62)
Bronchitis (Infections and infestations) | 0 | 4
Nasopharyngitis (Infections and infestations) | 2 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 4
Urinary Tract Infection (Infections and infestations) | 1 | 4
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 4
Headache (Nervous system disorders) | 3 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT06028438/Prot_002.pdf
  • Statistical Analysis Plan (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT06028438/SAP_003.pdf